CLINICAL TRIAL: NCT04870333
Title: PROphylaxis for paTiEnts at Risk of COVID-19 infecTion
Brief Title: PROphylaxis for paTiEnts at Risk of COVID-19 infecTion -V
Acronym: PROTECT-V
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Life Arc (Unknown); Kidney Research UK (KRUK) (Unknown); UNION therapeutics (Industry); Addenbrookes Charitable Trust (Other); GlaxoSmithKline (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr. Rona Smith, Senior Research Associate, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCTU0307; 2020-004144-28 (EudraCT Number)
Record Dates: First submitted 2021-03-01; First posted 2021-05-03 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Covid19
Keywords: dialysis; solid organ transplant; vasculitis; glomerulonephritis; systemic lupus erythematosus; haematopoietic stem cell transplant; oncology or haematology patient who is or has received chemotherapy or who is immunocompromised as a result of their disease or treatment; diagnosis of an autoimmune/inflammatory disease currently receiving immunosuppression; primary and secondary immunodeficiencies
MeSH Terms: conditions — COVID-19; Vasculitis; Glomerulonephritis; Lupus Erythematosus, Systemic; Neoplasms | interventions — Niclosamide; ciclesonide; sotrovimab

STUDY DESIGN:
Intervention Model Description: The following populations will be defined for efficacy and safety analyses:
  * Intent-to-treat population (ITT) The ITT population is defined as all participants randomised in the trial, regardless of whether they actually received trial treatment. The treatment group will be analysed as randomised.
  * Safety population The safety population comprises all participants randomised and having received as least one dose of trial treatment. The treatment group will be analysed as treated.
Who Masked: Participant, Care Provider, Investigator
Masking Description: PROTECT-V will be a double blind placebo controlled study where neither the participant nor clinician will be aware of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Niclosamide (Active Comparator): INN: Niclosamide Ethanolamine Chemical name (IUPAC): 5-chloro-N-(2-chloro-4-nitrophenyl)-2-hydroxybenzamide.2 aminoethanol CAS registry number: 1420-04-8 Lab code: UNI911
  The IMPs niclosamide Nasal Spray 1% and matching Nasal Spray Placebo will be provided in 20 mL amber glass vials with nasal spray pumps, containing 8.5 mL of the respective solution, delivering 140 μL per spray shot. It is an isotonic and euhydric aqueous solution with red colour.
  Interventions: Drug: Niclosamide
- Placebo niclosamide (Placebo Comparator): Placebo to match niclosamide will be supplied, stored, labelled, dispensed and dosed as for the active formulation. The placebo product is formulated to have the same appearance as the active solution.
  Interventions: Drug: Placebo
- Ciclesonide (Active Comparator): Chemical name (IUPAC): 2-[(1S,2S,4R,8S,9S,11S,12S,13R)-6-cyclohexyl-11-hydroxy-9,13-dimethyl-16-oxo-5,7-dioxapentacycloicosa-14, 17-dien-8-yl]- 2-oxoethyl 2-methylpropanoate CAS registry number: 141845-82-1
  It is a pressurised solution, intended for inhalation use and commercialised under the brand Alvesco. The recommended dose of ciclesonide is 160μg once daily, which leads to asthma control in the majority of patients. However, this may be increased if necessary to 320μg twice daily, in severe asthma.
  Interventions: Drug: Ciclesonide
- Placebo ciclesonide (Placebo Comparator): Matched placebo contains the same solvent and propellant as the active product but no drug substance.
  Interventions: Drug: Placebo
- Sotrovimab (Experimental): Sotrovimab, VIR-7831, GSK4182136 Sterile solution for intravenous infusion, 62.5 mg/mL, intravenous infusion Colourless or yellow to brown, liquid solution 20 mM histidine, 7% sucrose (w/v), 0.04% PS80 (w/v), 5 mM L-methionine at pH 6.0
  Interventions: Drug: Sotrovimab
- Placebo sotrovimab (Placebo Comparator): This will be in the form of 0.9% sodium chloride 100mL for infusion and will be sourced from commercially available stock by the site. It may be procured and stored as per sites usual procedures and only requires handling as an IMP upon dispensing and labelling.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide — 140μL of a 1% niclosamide ethanolamine solution in each nostril twice daily, equivalent to 1.4mg of niclosamide ethanolamine salt per nostril twice daily, approximately 12 hours apart. Total daily dose 5.6mg niclosamide ethanolamine salt (4.7mg free niclosamide acid). Treatment duration will be 6-9 months or up to 28 days after COVID-19 diagnosis unless hospitalised. Participants hospitalised with a diagnosis of COVID-19 should stop the randomised treatment immediately.
  Arms: Niclosamide
Drug: Placebo — 140μL of a matching placebo solution in each nostril twice daily. Treatment duration will be 6-9 months or up to 28 days after COVID-19 diagnosis unless hospitalised. Participants hospitalised with a diagnosis of COVID-19 should stop the randomised treatment immediately.
  Arms: Placebo niclosamide
Drug: Ciclesonide — Participants will be prescribed ciclesonide once daily, administered as follows:
  Two puffs (320 μg) inhaled via mouth sequentially One puff (160 μg) inhaled via nose Treatment duration will be 6-9 months or up to 28 days after COVID-19 diagnosis unless hospitalised. Participants hospitalised with a diagnosis of COVID-19 should stop the randomised treatment immediately.
  Arms: Ciclesonide
Drug: Placebo — Matched placebo: two puffs inhaled via mouth sequentially and one puff inhaled via nose.
  Treatment duration will be 6-9 months or up to 28 days after COVID-19 diagnosis unless hospitalised. Participants hospitalised with a diagnosis of COVID-19 should stop the randomised treatment immediately.
  Arms: Placebo ciclesonide
Drug: Sotrovimab — There will be a single infusion of sotrovimab administered at the beginning of the study.
  500mg of sotrovimab solution (8mL) will be diluted in 42mL of 0.9% sodium chloride and administered by intravenous infusion. 50mLs to be infused over 30 minutes with a 0.2 micrometre inline filter. Four vials will be required for a 2000 mg dose.
  Arms: Sotrovimab
Drug: Placebo — There will be a single infusion placebo, in the form of 100mL 0.9% sodium chloride, administered at the beginning of the study.
  Arms: Placebo sotrovimab

SUMMARY:
COVID-19 (SARS-CoV2 virus) was declared a global pandemic by the WHO on 11th March 2020. Currently there are no drugs proven to prevent COVID-19 or to reduce the severity of illness if given as prophylaxis. Although vaccines are now available, there remains a need for other prophylactic agents until vaccine use becomes widespread globally and effectiveness and durability is established, particularly in immunocompromised individuals, for whom vaccine responses may be suboptimal. Efforts are underway to repurpose established drugs with well understood drug interactions and safety profiles.

PROTECT-V is a platform trial to test prophylactic interventions against SARS-CoV2 infection in vulnerable patient populations at particularly high risk of COVID-19 and its complications, seeking to identify treatments that either might prevent the disease from occurring or may reduce the number of cases where the disease becomes serious or life-threatening.

In PROTECT-V, multiple agents can be evaluated on the same platform across vulnerable populations, with the option of adding additional treatments at later time points as these become available. The expectation is for as many sites as possible to recruit to all available trial treatments at any time, however, the platform structure and randomisation/data collection systems allow sites to open the trial treatment arms according to their capacity.

The trial opened with intranasal niclosamide and matched placebo, aiming to recruit 1500 vulnerable renal patients in February 2021. A parallel study protocol, was conducted in India, sponsored by The George Institute. Recruitment of around 750 Indian patients was completed in with the rest of the study arm recruitment in November 2022. The Niclosamide arm of the study was completed in June 2023.

The second agent, intranasal and inhaled ciclesonide and matched placebo, was meant to be added to the platform in mid-2022 in the same renal patient population however it was unable to be included due to other factor.

Sotrovimab and matched placebo have been added to the platform in August 2022 which aim to recruit approximately 800-1000 patients from the main study population with additional patient groups with primary immunodeficiency, any Haematology or Oncology patient who is currently receiving or has received chemotherapy or who is immunocompromised as a result of their disease or treatment, those with a diagnosis of an autoimmune or inflammatory disease receiving immunosuppression and also haematopoietic stem cell transplant recipients.

DETAILED DESCRIPTION:
Part 1: Inhaled repurposed agents The trial commenced with the first intervention, nasal niclosamide and matched placebo from February 2021. The intended second intervention is nasal and inhaled ciclesonide. Participants are being randomised in a 1:1 ratio until the second intervention is introduced. Once ciclesonide is introduced, participants who are eligible for ciclesonide will be randomised to niclosamide, ciclesonide, niclosamide matching placebo or ciclesonide matching placebo in a 2:2:1:1 ratio. The net result will be a 1:1:1 distribution between niclosamide, ciclesonide and placebo, with niclosamide-matching placebo and ciclesonide-matching placebo pooled for the analysis.

Three vulnerable patient populations were enrolled initially: dialysis patients, kidney transplant recipients and those with vasculitis or other auto-immune kidney disease such as systemic lupus erythematosus (SLE) or glomerulonephritis (GN) These patient groups are noted to be particularly vulnerable to COVID-19 infection by virtue of demographics, underlying co-morbidities or as a consequence of treatments for these conditions, and they are at exceptionally high risk of adverse outcomes. Additionally these groups are known to mount sub-optimal responses to vaccination.

Approximately 1500 participants will be randomised to active treatment or placebo, stratified by PROTECT sub-population, age and participating sites. Enrolment to the trial will be via an online platform following informed consent with a face to face screening visit. The screening visit will include assessment of eligibility (which will include liver function tests and COVID-19 PCR test), randomisation, baseline data collection and research serum sample collection to detect anti SARS-COV-2 antibodies. Subsequent assessments, aside from an in person end of trial visit, will be done via email or telephone together with utilising the routine collected health data thus reducing the burden to participants as well as reducing their exposure to COVID-19. Telephone consultations will be carried out at weeks 1, 2, 3, 4 and 6, followed by two weekly self-reporting at week 8 onwards.

If a participant has not submitted data for a period of approximately 6 weeks, they will be contacted by the local study team for a telephone interview to minimise loss to follow up. Failure to follow up a participant for more than 6 consecutive weeks will halt their trial treatment dispensation until communication has been restored. Failure to follow up a participant for more than 12 consecutive weeks will be considered loss of follow up and conclude their participation in the trial.

If a participant develops symptoms suggestive of COVID-19 infection they should arrange an urgent COVID-19 test. They should notify their trial physician. Participants should continue taking trial medication (if self-administering medication) until advised to stop by a member of the trial team or admitted to hospital. Any participant testing positive for SARS-CoV-2 will be required to complete a COVID-19 symptom assessment at least weekly for 4 weeks after diagnosis, unless hospitalised.

A final safety assessment will be conducted in person, 4-6 weeks after the final treatment. Participants will be asked to return all completed medication diaries and IMP containers, if self-administering, for compliance assessment at this visit. Participants will be asked a series of questions to identify any additional adverse events or adverse reactions experienced since their last follow up assessment and a blood sample will be taken for a SARS-CoV2 total antibody assay, to detect asymptomatic cases of COVID-19 infection. At the final assessment, patients may be re-screened for consideration of enrolment into one of the other arms of the PROTECT-V trial platform. It is not permitted for re-enrolment into the originally assigned arm.

Participants will continue allocated treatment until one of the following occurs:

1. The required number of the primary outcome events have occurred (for each intervention)
2. The participant is hospitalised with COVID-19 (see 4.10.2.)
3. 28 Days after a diagnosis of COVID-19 if hospitalisation is not required

The anticipated median treatment duration per participant is 6 months. However, the individual arm may conclude while some participants are in the trial for less than 6 months if the required number of events are observed. All Adverse Events and Adverse Reactions will be recorded in the medical notes and in the appropriate section of the case report form. Serious adverse events and serious adverse reactions should be reported to the sponsor.

Niclosamide is a derivative of salicylic acid and has been used to treat tapeworm infections. The exact target and mechanism of action is uncertain. Researchers at Institut Pasteur Korea have reported niclosamide as one of the most potent FDA approved inhibitors of SARS-Cov-2 in in vitro assays using vero cells, with IC50 of 0.28μM >25x higher than that of chloroquine and >40x higher than that of remdesivir. In-vitro data indicating potent inhibition of SARS-COV2 replication and cellular penetration, together with evidence that SARS-COV2 initially replicates predominantly in the nasal epithelium, suggests nasal niclosamide is best placed as a prophylactic agent or for treatment of early stage COVID-19 disease when the viral load is a main issue. Hepatic clearance is the primary mechanism for elimination and there is anticipated low bioavailability, therefore no dose adjustments are required for patients with renal impairment. Side-effects (based on a phase 1 study in healthy volunteers) are minor nasal irritation, sneezing or runny nose. Population Pharmacokinetic (PK) assessment will be conducted in the first 30 participants receiving niclosamide for safety purposes, to exclude the unlikely possibility of accumulation of niclosamide during the course of the trial in patients receiving dialysis only.

Ciclesonide is an inhaled corticosteroid (ICS) that has been shown to possess in vitro anti-SARS-CoV-2 activity. Ciclesonide inhibits in vitro SARS-CoV-2 replication in cultured human bronchial epithelial cells via a novel mechanism on non-structural protein 15 (NSP-15). ICS, particularly at higher doses, have been shown to reduce expression of ACE2 and TMPRSS2 receptors, which mediate infection of host respiratory epithelial cells. ICS have also been shown to inhibit in vivo production of IL-6, a key pro-inflammatory cytokine in COVID-19 and a major predictor of severe disease and poor outcomes. The proposed combination of prophylactic inhaled and intranasal ciclesonide will deliver early infection modifying therapy covering the entire respiratory epithelium, critical in the early stages of COVID-19. Ciclesonide and its active metabolite are metabolised and excreted by hepatic mechanisms, therefore no dose adjustments are required for patients with renal impairment, Side-effects may include cough, bronchospasm, bad taste and application site reactions.

Part 2: Monoclonal antibodies and anti-viral agents

Sotrovimab is a fully human IgG1κ monoclonal antibody (mAb) derived from the parental mAb S309, a potent neutralising mAb directed against the spike protein of SARS-CoV-2. S309 binds to a highly conserved epitope of the SARS-CoV and SARS-CoV-2 spike protein receptor binding domain (RBD) and inhibits SARS-CoV-2 infection in vitro. Sotrovimab demonstrates high affinity binding to the SARS-CoV-2 spike RBD. COMET-ICE is a Phase II/III randomised, double-blind, placebo-controlled study which evaluated sotrovimab as treatment for COVID-19 infection in non-hospitalised patients at high risk of medical complications of the disease. The primary endpoint, progression of COVID-19 at Day 29, was reduced by 85% compared with placebo.

A single dose of 500 mg was selected for the study based on in vitro neutralisation data, in vitro resistance data, and IV PK data from the COMET-ICE [NCT04545060] study. No dose modification is required in renal or hepatic disease. The overall rate of AEs in COMET-ICE was similar in those treated with sotrovimab compared to placebo. The known side-effects of sotrovimab are hypersensitivity and anaphylaxis. There will be a single infusion of sotrovimab or placebo administered at the beginning of the study. Based on the pharmacokinetics of the drug, it is predicted that the single infusion will remain efficacious for approximately 16 weeks.

An absent or suboptimal response (Roche Elecsys® Anti-SARS-CoV-2 assay result <400 AU/mL) to COVID-19 vaccination, assessed at least 14 days after the vaccine was initially require to be eligible for the sotrovimab arm of the study however, this have been remove from the criteria. Additional patient groups with primary immunodeficiency, any Haematology or Oncology patient who is currently receiving or has received chemotherapy or who is immunocompromised as a result of their disease or treatment, those with a diagnosis of an autoimmune or inflammatory disease receiving immunosuppression and also haematopoietic stem cell transplant recipients have been added.

In addition to the core components of the screening visit previously listed the following will also be conducted: ECG, serum antibody sample for Roche Elecsys® Anti-SARS-CoV-2 assay, full blood count, clotting profile, renal and liver function test (routine ALT/AST tests performed up to 2 week before screening visit will be accepted to assess liver function), and serum pregnancy test in women of child bearing potential, urine albumin: creatinine ratio.

At the day 1 infusion visit, prior to commencing the IMP infusion, a blood sample to measure anti-drug antibodies will be collected. Routine observations must be taken prior to infusion, at the end of infusion and 1 hour after infusion and to be recorded. PK samples to be taken within 1 hour after end of infusion.

Telephone consultations/remote telephone assessments will be carried out weekly for the first 4 weeks, alternative weeks from week 6 to 24 and then every 4th week from week 28 to 36. In person assessments will occur during weeks 4, 12 and 24 and will include blood sample collection for measurement of COVID-19 antibodies and PK sampling.

ELIGIBILITY:
Core protocol

Inclusion Criteria:

* Be aged 18 years or older
* Have given written informed consent
* Be a member of one of the following vulnerable patients populations

  * Dialysis - including in centre haemodialysis, home haemodialysis and peritoneal dialysis
  * Kidney transplant receiving at least one of the immunosuppressive medications listed below
  * Vasculitis (according to Chapel Hill Consensus Conference 2012 definitions) or systemic lupus erythematosus (SLE) receiving at least one of the immunosuppressive medications listed below
  * Glomerulonephritis (includes prior histological confirmation of any of the following conditions - minimal change nephropathy, focal segmental glomerulosclerosis (FSGS), IgA nephropathy, primary membranous nephropathy, membranoproliferative glomerulonephritis or lupus nephritis) receiving at least one of the immunosuppressive medications listed below Ciclosporin Tacrolimus Azathioprine Mycophenolate Mofetil or Mycophenolic Acid Belatacept Methotrexate Tocilizumab Abatacept Leflunomide Sirolimus Prednisolone (current dose) > 20mg daily for 8 weeks Anti-TNF (infliximab, adalimumab, etanercept) Belimumab Cyclophosphamide (within the last 6 months) Rituximab (in the last 12 months) or Rituximab in the last 5 years and IgG level <5g/l Alemtuzumab (in the last 12 months)

Exclusion Criteria:

* Inability to provide informed consent or to comply with trial procedures
* COVID-19 at time of enrolment - either positive SARS CoV-2 swab (PCR) or symptoms highly suggestive of COVID-19 infection
* Known chronic liver disease or hepatic dysfunction as evidenced by ALT or AST > 3x upper limit of the normal range
* Allergy or hypersensitivity to any of the active IMPs, or to any of the excipients used
* Pregnant, trying to conceive, unwilling to use contraception or breastfeeding
* Current participation in another interventional prophylactic or vaccine trial* against COVID-19.

  * Patients remain eligible for enrolment if they have received SARS-COV-2 vaccination as part of routine care.

NICLOSAMIDE ARM Additional exclusion criteria

* Significant structural nasal disease in the opinion of the investigator
* Prior participation in the niclosamide arm of the trial (if being re-screened for participation in a second interventional arm).

CICLESONIDE ARM Additional Exclusion Criteria

In addition to the core exclusion criteria in the master protocol, the presence of any of the following will preclude participant inclusion:

1. Significant structural nasal disease in the opinion of the investigator
2. Prior participation in the ciclesonide arm of the trial (if being re-screened for participation in a second interventional arm).
3. Currently taking inhaled corticosteroids - beclometasone dipropionate (aerosol inhaler and dry powder inhaler), budesonide (dry powder inhaler and single-dose units for nebulization), ciclesonide (aerosol inhaler), fluticasone propionate (dry powder inhaler, aerosol inhaler, and single-dose units for nebulization), mometasone furoate (dry powder inhaler).
4. Received a live vaccine within last 14 days - ciclesonide increases risk of generalised infection: influenza, MMR, rotavirus, typhoid, varicella-zoster (shingles), yellow fever.
5. Taking one of the following medications ○ Systemic Ketoconazole, itraconazole, ritanovir, nelfinavir

SOTROVIMAB ARM Additional Inclusion Criteria

• Be a member of an immunocompromised population, which includes but is not limited to those groups listed in the core protocol as well as the following:

* Primary immunodeficiency
* Any Oncology, Haematology-Oncology or Haematology patient who is currently receiving or has received chemotherapy or who is immunocompromised as a result of their disease or treatment
* Have a diagnosis of an autoimmune/inflammatory disease currently receiving immunosuppression including those individuals currently on Prednisolone ≥20mg daily for at least 4 weeks. Those who have received Rituximab or Alemtuzumab within the last 12 months would also be eligible.
* Solid organ and haematopoietic stem cell transplant recipients

Additional Exclusion Criteria

In addition to the core exclusion criteria in the master protocol, the presence of any of the following will preclude participant inclusion:

* If in the opinion of the PI it is not in the best interests of the participant to take part in the study - for example due to limited life expectancy (≤12 months) due to pre-existing co-morbidities
* History of hypersensitivity reaction to sotrovimab, one of its excipients or any other monoclonal antibody targeting SARS CoV-2
* History of receiving any monoclonal antibody targeting SARS CoV-2 within the last 6 months
* Admission to hospital for acute, unplanned care at the time of randomisation or in the two weeks prior to screening
* History of receiving chimeric antigen receptor T-cell (CAR-T) therapy less than 4 weeks prior to consenting to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2240 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Confirmed symptomatic COVID-19 infection during treatment | 6-9 months. Reported at 24 weeks for niclosamide and ciclesonide arms and 12 weeks for sotrovimab arm from date of IMP administration.
  The primary outcome for PROTECT is confirmed symptomatic COVID-19 infection during treatment.
  The primary outcome event is defined as the presence of both
  * PCR confirmed SARS-CoV2 and
  * One or more symptoms in keeping with COVID-19, including:
    * Respiratory (Cough +/- sputum and shortness of breath)
    * Constitutional (Pyrexia/chills, myalgia/arthralgia, fatigue, rash, headache, confusion)
    * Gastrointestinal (nausea/vomiting, diarrhoea, abdominal pain, loss of appetite) The date (time) of the primary outcome event is defined as the date of the confirmed COVID-19 test.

SECONDARY OUTCOMES:
Time to confirmed SARS-Cov-2 infection from the date of randomisation including asymptomatic cases. In addition, confirmed symptomatic COVID-19 infection at 16, 24, 36, and 48 weeks from date of IMP administration. | 6-9 months
Safety and seriousness of the event | 9 months
  SAE and SAR since consent until end of follow-up or at the time of withdrawal from the study. Safety will be assessed weekly for the first 4 weeks and then 2-weekly from 6th week onwards using a questionnaire that includes common COVID symptoms and all expected reactions to the trial. Investigators will also report any SAE or SAR within 24 hours of awareness.
All-cause mortality | 9 months
Severity of COVID-19 disease | 28 days after date of positive test
  Severity of COVID-19 disease (assessed by PI 28 days after date of positive test following current guidelines)

OTHER OUTCOMES:
Occurrence of other infections | 6-9 months
  Occurrence of other influenza infection (swab confirmed) - niclosamide arm only Occurrence of other respiratory viral infections (aside from COVID-19 and influenza) Staphylococcus aureus infections (dialysis population only)

CONTACTS AND LOCATIONS:
Overall Officials: Rona Smith, Dr, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (45):
- United Kingdom (45):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - NHS Lanarkshire - University Hospital Monklands, Airdrie
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Betsi Cadwaladr University Health Board, Bodelwyddan
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - North Bristol NHS Trust, Bristol
  - West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Cardiff & Vale University Health Board, Cardiff
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton
  - Ayrshire & Arran NHS Trust, Crosshouse
  - Dartford and Gravesham NHS Trust, Dartford
  - University Hospitals of Derby and Burton NHS Trust, Derby
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - NHS Tayside, Dundee
  - The Royal Devon and Exeter NHS Foundation Trust, Exeter
  - James Paget University Hospital NHS Foundation Trust, Great Yarmouth
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Queen Elizabeth Hospital, King's Lynn, NHS Foundation Trust, Kings Lynn
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Royal Free NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Royal Berkshire NHS Foundation, Reading
  - Salford Royal NHS Foundation, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - The Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - East and North Hertfordshire NHS Trust, Stevenage
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland
  - The Royal Wolverhampton NHS Trust, Wolverhampton
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data meta-analysis that underlie the results reported in this article would be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication and after 36 months the data will be available in our University's data warehouse however without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at the link below
URL: https://www.camcovidtrials.net/trials/protect.htm

REFERENCES:
- [Derived] Humphrey TJL, Qian W, Chen-Xu M, Dowling F, Gatley K, Adhikari R, Hensman T, Stockley L, Bassi A, Bathla N, Dasgupta I, Dosanjh DPS, Jellingso M, Sorensen P, Jensen ML, Callesen AW, Bradley JR, Jha V, Sommer MOA, Hiemstra TF, Smith RM; PROTECT-V consortium. Prophylaxis for renal patients at risk of COVID-19 infection: results from the intranasal niclosamide randomised, double blinded, placebo controlled arm of the PROTECT-V platform trial. BMC Infect Dis. 2025 Feb 11;25(1):204. doi: 10.1186/s12879-025-10584-4. PMID 39934669
- [Derived] Humphrey TJL, Dosanjh D, Hiemstra TF, Richter A, Chen-Xu M, Qian W, Jha V, Gatley K, Adhikari R, Dowling F, Smith RM. PROphylaxis for paTiEnts at risk of COVID-19 infecTion (PROTECT-V). Trials. 2023 Mar 13;24(1):185. doi: 10.1186/s13063-023-07128-z. PMID 36915199
- See also: PROTECT website — https://www.camcovidtrials.net/trials/view,protect_50.htm

DOCUMENTS (1):
  • Study Protocol (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT04870333/Prot_001.pdf